CLINICAL TRIAL: NCT05285748
Title: Comparing a Recommendation for Self-paced Versus Moderate Intensity Physical Activity for Midlife Adults: an RCT
Brief Title: Comparing Self-paced Versus Moderate Intensity Physical Activity Recommendation for Midlife Adults
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, David M. Williams, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R01AG069349 (NIH); F32AG074680 (NIH)
Record Dates: First submitted 2022-02-23; First posted 2022-03-18 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Physical Inactivity
Keywords: Physical activity; Exercise; Self-pacing
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Paced Intensity Physical Activity (Experimental)
  Interventions: Behavioral: Self-Paced Intensity Physical Activity
- Prescribed Moderate Intensity Physical Activity (Active Comparator)
  Interventions: Behavioral: Prescribed Moderate Intensity Physical Activity

INTERVENTIONS:
Behavioral: Self-Paced Intensity Physical Activity — Participants are given a prescription to engage in 150-300 minutes per week of structured exercise with an emphasis on walking. For this study arm, participants are given the explicit recommendation to engage in self-selected intensity PA.
  Arms: Self-Paced Intensity Physical Activity
Behavioral: Prescribed Moderate Intensity Physical Activity — Participants are given a prescription to engage in 150-300 minutes per week of structured exercise with an emphasis on walking. For this study arm, participants are given the explicit recommendation to engage in moderate intensity PA consistent with national guidelines.
  Arms: Prescribed Moderate Intensity Physical Activity

SUMMARY:
We will randomly assign (blocked on Gender (female, male, other), body mass index (BMI; overweight [25 < BMI < 30]) or obese (30 < BMI <40) and pain status (chronic pain vs not)) adults ages 50-64 into either; (a) self-selected intensity (i.e., SELF-PACED) or (b) prescribed moderate intensity (i.e., PRESCRIBED) conditions. Prior to randomization, persons responding to our ads will participate in the following: (1) telephone screening with the study research assistant (RA) to establish eligibility; (2) an orientation session to obtain more information about the study; and, after providing informed consent (3) baseline assessment and screening (bodyweight, maximal fitness test, dietary intake, and questionnaires to assess potential covariates). Prior to randomization, the RA will give participants an accelerometer to assess baseline physical activity (PA) behavior over a one-week period. Participants will then be randomized to one of the two study conditions. Following randomization, all participants will receive our theory-based PA promotion intervention to help them overcome barriers to regular PA. All participants will be given chest strap heart rate (HR) monitors and instructions on wrist palpation. Follow-up assessments will consist of accelerometry for one-week periods at months 3, 6, 9, and 12, ecological momentary assessment (EMA) throughout the 12 months and bodyweight at 3-month intervals.

ELIGIBILITY:
Inclusion criteria:

* ages 50-64
* BMI 25-40
* Sedentary or low-active, defined as participating in < 60 min/week of structured exercise
* Has a smart phone that can connect to the internet at least once every few days and is compatible with smartphone app

Exclusion criteria:

* Medical symptoms/conditions that may make unsupervised exercise unsafe (specific exclusion criteria were developed in consultation with a cardiologist and are listed below):

  * Past 3-month overnight hospitalization
  * Past 3-month treatment for heart disease, including bypass or valve surgery, interventional procedure(s) such as angioplasty (stent), or a pacemaker or other implanted device to control your heart rate or rhythm
  * Past 3-month inability to walk without assistance due to stroke, transient ischemic attack (TIA), or neurologic or spinal injury
  * Past 6-month angina, chest pain, or chest discomfort either at rest or with exertion/activity
  * Past 6-month peripheral vascular disease such as claudication which causes pain in the legs when walking briskly
  * Past 6-month seizure
  * Past 6-month overnight hospitalization due to respiratory disease
  * Past 6-month lightheadedness, vertigo, dizziness, or fainting
  * Heart, lung, abdominal, joint, or orthopedic surgeries in the past 12-months, or pending or scheduled in the next 12 months
  * Takes insulin and/or medication that affects the secretion of insulin
  * Exercise-induced asthma that prevents brisk walking
  * Takes anticonvulsant medication or medication to treat/control seizures
  * Diagnosed with cystic fibrosis
  * Bone or joint problems that make you unable to walk for at least 30 minutes
  * Physician has said not to exercise because of bone or joint problems
  * Physician has said a hip or knee replacement will be needed in the next 12 months
  * Anything other medical symptoms/condition that prevents participant from being physical unable to walk without assistance continuously for 30 minutes
* Currently taking or planning on taking medications that affect HR, such as beta or calcium channel blockers or digoxin, as HR will be used to determine the moderate intensity range for participants assigned to that condition
* Past 12-month overnight psychiatric hospitalization
* Currently pregnant or planning to become pregnant in the next year
* Currently participating in any exercise or weight-loss research studies
* Household member is participating in this study
* Does not have a Rhode Island mailing address OR if only Rhode Island mailing address is a PO box
* Unable to receive materials in the mail at residential mailing address
* Does not plan to live in Rhode Island for the next 12 months
* Unable to speak, read, and/or write fluently in English
* Smokers will be eligible, but smoking status will be included as a covariate in analyses

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 258 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in total volume of structured PA | Measured at baseline, and months 3, 6, 9, and 12.
  Minutes of PA weighted by intensity, expressed in metabolic equivalent (MET) minutes as determined by accelerometers (Actigraph [model wGT3x-BT]) worn during one-week periods.
Minutes per week of PA | Measured daily from date of randomization for 52 weeks based on participant initiation of exercise
  Participants will be instructed to indicate, in real time, each time they begin and end a PA session via EMA.

SECONDARY OUTCOMES:
Changes in Body Weight | Measured at baseline, and months 3, 6, 9, and 12.
  Assessment of self-reported body weight by study-provided scales

OTHER OUTCOMES:
Opportunity Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's opportunity to do regular aerobic physical activity
Capability Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's physical and psychological capability to do regular aerobic physical activity
Exercise Motivation Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's motivation on the days they have made a plan to exercise
Habit of Physical Activity Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's habits regarding exercise
Physical Activity Identity Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's personal beliefs regarding exercise
Outcome Expectations for Physical Activity Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's beliefs about the consequences of exercise
Attitude towards Physical Activity - Affective Attitude Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's beliefs about exercise
Attitude towards Physical Activity - Instrumental Attitude Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's beliefs about exercise
Physical Activity Enjoyment Scale (title of questionnaire; not subscale; measuring changes in PA enjoyment) | Measured at baseline, and months 3, 6, 9, and 12.
  Measures how much a person enjoys exercise; scores range from 18-26 and higher scores mean more physical activity enjoyment
Intention Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's intention to exercise
Chronic Pain Screening Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures how much chronic pain a person had in the past 6 months
Pain Medication Use Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures the medications a person is taking for chronic pain
12 Item Short Form (SF-12) Health Survey | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's views about their health
Quality of Life Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's views about their quality of life and health
Activity Tracker Use Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures of use of physical activity devices, memberships, and equipment
EMA: Affective response to PA | Upon participant initiation of PA session, measured before, during, and after PA sessions; beginning at randomization through 52 weeks of study
  Captures the shift in core affective valence (feeling good vs bad) from pre-PA to during-PA.
EMA: Perceived autonomy | Measured weekly from date of randomization until the end of the study at week 52
  Assesses participant's perceived autonomy over exercise behavior.
EMA: Perceived exertion | Measured daily from date of randomization until the end of the study at week 52
  Assesses participant's perceived exertion during PA.
EMA: Behavioral intention | Measured daily from date of randomization until the end of the study at week 52
  Assesses degree to which participant intends to engage in PA.
EMA: PA setting | Measured daily from date of randomization until the end of the study at week 52
  Assessed the physical and social setting in which a participant engages in physical activity.
EMA: Anticipated, remembered, and incidental affect | Measured daily from date of randomization until the end of the study at week 52
  Will assess how participant expects to feel after engaging in PA, how participant remembers feeling after engaging in PA, and how participant currently feels.
EMA: Self-Efficacy for Physical Activity | Measured daily from date of randomization until the end of the study at week 52
  Measures beliefs about capabilities to be physically active
EMA: Social Support for Exercise | Measured daily from date of randomization until the end of the study at week 52
  Measures a person's social support available to help them exercise

CONTACTS AND LOCATIONS:
Overall Officials: David M Williams, Ph.D., Principal Investigator — Brown University School of Public Health
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT05285748/ICF_000.pdf